CLINICAL TRIAL: NCT01133171
Title: A Personalized Dashboard to Educate Veterans at Risk of Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 09-186
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Cardiovascular Disease; Stroke
Keywords: Cardiovascular Disease; Stroke
MeSH Terms: conditions — Cardiovascular Diseases; Stroke | interventions — Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dashboard Plus Nurse (Experimental): Patients randomized to this intervention arm were seen twice over six months by a research nurse to collect data on risk factors and received counseling plus a computerized dashboard intervention.
  Interventions: Behavioral: Nurse Alone; Behavioral: Dashboard Plus Nurse
- Nurse Alone (Experimental): Patients randomized to this intervention arm were seen twice over six months by a research nurse to collect data on risk factors and received counseling.
  Interventions: Behavioral: Nurse Alone
- Control (No Intervention): Patients randomized to this group were followed retrospectively to collect data on their primary care visits and laboratory results and past medical history over the 12 month study period. They had no contact with study personnel and did not receive any type of intervention.

INTERVENTIONS:
Behavioral: Nurse Alone — Patients received two in-person counseling sessions by a research nurse, approximately 3-7 months apart, in methods for controlling cardiovascular risk factors.
  Arms: Dashboard Plus Nurse; Nurse Alone
Behavioral: Dashboard Plus Nurse — Patients receive two in-person counseling sessions, six months apart, in methods for controlling cardiovascular risk factors and were asked to use a computerized dashboard to enter values for the risk factors and observe the effects of the risk factors on the overall cardiovascular risk.
  Arms: Dashboard Plus Nurse

SUMMARY:
Personalized risk communication methods have been used to educate patients that are at a high risk of developing cardiovascular disease. These methods include personalized counseling, printed brochures and individualized graphs describing the status of the risk factors. Very few studies have provided an interactive tool for patients to self-manage their risk factors and observe the changes in risk by making lifestyle changes and modifying other risk factors by seeking medical advice.

This Rapid Response Project (RRP) builds upon these methods of communication by presenting the modifiable risk factors in the form of a personalized dashboard that highlights the contribution of these risk factors on the risk of developing a cardiovascular event. The modifiable risk factors that will be addressed in this study will include medical and lifestyle risk factors. The medical risk factors are hypertension, atrial fibrillation, diabetes mellitus and hyperlipidemia whereas the lifestyle risk factor is tobacco use.

Our primary goal is to develop a prototype of the dashboard to educate patients and help them make informed decisions in modifying their risk factors to reduce the probability of a cardiovascular event or stroke. We will also evaluate the effectiveness of this tool by asking these patients to return after 6 months to determine if they have made any lifestyle changes or pursued medical intervention to reduce their cardiovascular risk. We will make qualitative observations on the knowledge retention of these patients while using the interactive dashboard.

DETAILED DESCRIPTION:
Background:

Personalized risk communication methods have been used to educate patients who are at high risk of developing a cardiovascular event. These methods include personalized counseling, printed brochures and individualized graphs describing the status of the risk factors. Very few studies have provided an interactive tool for patients to use to compare the relative change in risk that might result from modifying their risk factors.

Objectives:

The goals of this pilot study were to: (a) develop a prototype of a personalized dynamic dashboard to educate veterans and help them make informed decisions about modifying their vascular risk factors (hypertension, diabetes mellitus, hyperlipidemia, and tobacco use) to reduce the probability of a vascular event; (b) test the usability of this tool from the patient's perspective; and (c) provide preliminary data regarding the effectiveness of this tool in terms of changes in lifestyle or risk factor control compared with nurse-education.

Methods:

This was a three-arm randomized controlled study. Veterans from the panel of one experienced general internist were randomly assigned to one of three groups: (1) dashboard with nurse-education, (2) nurse-education alone, (3) usual care. To be eligible, patients must have had at least two of the following: body mass index >30 kg/m2; current tobacco use; systolic blood pressure >140 mm Hg or diastolic >90 mm Hg; LDL-cholesterol >130 mg/dL, or hemoglobin Hb1Ac >8%. We developed the dashboard in our Human Computer Interface/Information Technology laboratory. Patients in the dashboard group received two in-person counseling sessions regarding methods for controlling risk factors, and were asked to use the dashboard tool to enter values for their own risk factors and to observe the relative effects of varying their risk factor control on their overall vascular risk. The nurse-education consisted of two in-person counseling sessions regarding methods for controlling risk factors. Both intervention sessions lasted approximately 30 minutes; therefore, the majority of the time was used to interact with the tool in the dashboard group whereas the entire time was used for personalized risk factor discussion in the nurse-education group. For the usual care group, data were retrospectively collected about the primary care visits and laboratory tests which took place during the same period as the visits for intervention patients.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving care from a Primary Care Clinic at the Roudebush VA Medical Center in Indianapolis with at least two of the following risk factors:
* Body Mass Index > 30
* Current Smoker
* Systolic Blood Pressure > 140 mm OR Diastolic Blood Pressure >90 mm
* Cholesterol LDL > 130 mg/dL
* Hemoglobin Hb1Ac > 8%

Exclusion Criteria:

* Subjects on Dialysis
* Subjects on Supplemental Oxygen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Merchant, PhD MSc, Principal Investigator — Richard Roudebush VA Medical Center, Indianapolis
Locations (1):
- Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dashboard Plus Nurse | Nurse Alone | Control
Started | 25 | 27 | 25
Completed | 24 | 25 | 25
Not Completed | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dashboard Plus Nurse | Nurse Alone | Control | Total
Number analyzed (Participants) | 24 | 25 | 25 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.2) | 61.9 (12.5) | 62.8 (10.5) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 23 | 25 | 25 | 73
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 25 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Participants Who Initiate Conversation With Primary Care Provider About Vascular Risk
Description: Only the intervention patients were analyzed for this outcome.
Time Frame: From baseline to six-months
Measure: Number; unit: percentage of patients
Arm/Group | Dashboard Plus Nurse | Nurse Alone
Number analyzed (Participants) | 24 | 25
percentage of patients | 11.1 | -21.4

2. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: From baseline to six months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dashboard Plus Nurse | Nurse Alone | Control
Number analyzed (Participants) | 24 | 25 | 25
mmHg | -0.8 (18.1) | -2.3 (11.3) | 8.4 (19.1)

ADVERSE EVENTS:
Time Frame: The six-month period
Arm/Group | Dashboard Plus Nurse | Nurse Alone | Control
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes